CLINICAL TRIAL: NCT01559688
Title: Accelerated Resolution Therapy (ART) for Psychological Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TATRC-01
Record Dates: First submitted 2011-10-19; First posted 2012-03-21 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2013-10

CONDITIONS: Psychological Trauma; PTSD
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ART therapy group (Experimental): Participants in this arm will receive 2-5 sessions of ART therapy, depending on individual progress. Each session will last 60-90 minutes over a 2-week period.
  Interventions: Behavioral: Accelerated Resolution Therapy (ART)
- Waitlist (Active Comparator): Participants in this group will receive 2 fitness assessment or career counseling sessions. Each session will last 60-90 minutes over a 2-week period. Upon completion of this arm, participants will be offered the choice to start ART therapy.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Accelerated Resolution Therapy (ART) — ART is a cognitive based therapy which integrates an eye movement technique while focusing on a problem (traumatic experience) during the therapy session.
  Arms: ART therapy group
Behavioral: Waitlist — Fitness assessment or career counseling
  Arms: Waitlist

SUMMARY:
Service members and veterans often experience symptoms of psychological trauma following combat deployments. While efforts are being made in the military and at the Veteran's Affairs to meet the large number of soldiers and veterans experiencing symptoms of psychological trauma, there remains a need to evaluate new treatments, particularly those that are designed to be brief in length.

A new therapy, known as Accelerated Resolution Therapy (ART), is a type of psychological therapy that is designed for rapid resolution of symptoms of psychological trauma. This approach uses a combination of talking and sets of eye movements guided by the therapist. During therapy, this interactive personal guidance is thought to be helpful in resolving problems (such as bad memories).

The purpose of this study is to:

1. Evaluate how effective ART is in treating symptoms of psychological trauma among non-active duty veterans who served in Operation Iraqi Freedom and Operation Enduring Freedom in Iraq and in Afghanistan or other combat conflicts.
2. Learn if there is improvement in symptoms of psychological trauma (such as bad memories, anxiety, depression, and guilt) after receiving Accelerated Resolution Therapy (ART).

ELIGIBILITY:
Inclusion Criteria:

* Non-active duty U.S. veteran of any prior deployment(s) with recruitment emphasis on those who previously served in Iraq and/or Afghanistan (OIF and OEF).
* At least 18 years of age.
* Symptoms indicative of psychological trauma. This includes a score of >40 on the PCL-M Checklist, or in the absence of a score >40, therapist assessment of symptoms of PTSD, as determined from the Checklist for Accelerated Resolution Therapy (ART) Standard Protocol. Individuals with previous treatment for psychological trauma, yet with residual symptoms, will be eligible.
* Ability to read and speak English to complete survey questions.
* Denial of suicidal ideation or intent, including homicidal ideation or intent, and no evidence of psychotic behavior or being in psychological crisis

Exclusion Criteria:

* Brain injury prohibiting speech, writing, and purposeful actions
* Identified to have current suicidal ideation
* Major psychiatric disorder concomitant to symptoms of psychological trauma
* Currently undergoing substance abuse treatment
* Previous diagnosis of eye movement disorder
* Any medical condition that, in the judgment of the Principal Investigator and/or ART therapist, may place the individual at high risk due to a potential heightened emotional reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Checklist (PCL-M) score from baseline to end of treatment | approximately 2 weeks
  This questionnaire asks about symptoms in response to "stressful military experiences."

SECONDARY OUTCOMES:
Change in psychological wellness as measured by Brief Symptom Inventory from baseline to endpoint | approximately 2 weeks
Change in trauma-related guilt as measured by Trauma-Related Guilt Inventory from baseline to endpoint | approximately 2 weeks
Change in depressive symptoms as measured by the Center for Epidemiologic Depression (CES-D) scale from baseline to endpoint | approximately 2 weeks
Change in anxiety symptoms as measured by State-Trait Inventory from baseline to endpoint | approximately 2 weeks
Change in anger as measured by Aggression Questionnaire from baseline to endpoint | approximately 2 weeks
Change in sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI) from baseline to endpoint | approximately 2 weeks
Change in self-compassion scale score from baseline to endpoint | approximately 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kip, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Kip KE, Shuman A, Hernandez DF, Diamond DM, Rosenzweig L. Case report and theoretical description of accelerated resolution therapy (ART) for military-related post-traumatic stress disorder. Mil Med. 2014 Jan;179(1):31-7. doi: 10.7205/MILMED-D-13-00229. PMID 24402982
- [Derived] Kip KE, Rosenzweig L, Hernandez DF, Shuman A, Sullivan KL, Long CJ, Taylor J, McGhee S, Girling SA, Wittenberg T, Sahebzamani FM, Lengacher CA, Kadel R, Diamond DM. Randomized controlled trial of accelerated resolution therapy (ART) for symptoms of combat-related post-traumatic stress disorder (PTSD). Mil Med. 2013 Dec;178(12):1298-309. doi: 10.7205/MILMED-D-13-00298. PMID 24306011